CLINICAL TRIAL: NCT02446379
Title: Evaluation of the Use of Intra-operative Molecular Imaging With BetaScope and in Vitro Measurement With LightPath Specimen Analyser Devices in Gastrointestinal Tumour Surgery
Brief Title: Use of the EnLightTM and LightPathTM Imaging Systems in Gastrointestinal Tumour Surgery
Acronym: CLIO
Status: Withdrawn | Type: Observational
Why Stopped: Technology licensed to third party. Sponsor did not proceed with study.
Sponsor: Lightpoint Medical Limited (Industry)
Collaborators: Semmelweis University (Other)
Responsible Party: Sponsor
Other Study IDs: LPM-005
Record Dates: First submitted 2015-04-27; First posted 2015-05-18 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Gastric Cancer; Pancreatic Cancer; Bile Duct Cancer; Duodenal Cancer
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms; Bile Duct Neoplasms; Duodenal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EnLightTM and LightPathTM Imaging Systems arm: Patients will first be injected intravenously with 2-5 MBq/kg, up to a maximum 300 MBq of the marketed product 18F-fluorodeoxyglucose (FDG) and after this undergo tumour excision surgery according to standard of care.
  The surgical cavity will be imaged by the EnLightTM system and the tumour excision specimen will be imaged by both the EnLightTM and LightPathTM Imaging Systems. The EnLightTM and LightPathTM Imaging Systems results will not influence any surgical or clinical decision-making. The tumour excision specimen will be analysed according to standard of care pathology. Patients will be followed-up (Visit 3) 2-14 days after the end of surgery for adverse events (AEs).
  Interventions: Drug: The marketed product 2-5 MBq/kg 18F-fluorodeoxyglucose; Device: EnLightTM; Device: LightPathTM Imaging System

INTERVENTIONS:
Drug: The marketed product 2-5 MBq/kg 18F-fluorodeoxyglucose — The FDG is injected at least 120 minutes prior to the imaging by the EnLightTM and LightPathTM Imaging Systems
  Other Names: FDG
Device: EnLightTM — The surgical cavity and the resected lymph nodes (if any) will be imaged by the EnLightTM system to establish whether radioactive tissue remains after surgery.
Device: LightPathTM Imaging System — The resected tumour excision specimens and the resected lymph nodes (if any)will be imaged by CLI and by WLI to establish whether they contain radioactive tissue.

SUMMARY:
This study will evaluate the performance of the EnLightTM and LightPathTM Imaging Systems in detecting tumour lesions in patients with gastric, pancreas, bile duct or duodenal cancer.

EnLightTM will be used to detect positron emission and the LightPathTM system to detect Cerenkov Luminescence. Both are emitted by the Positron Emission Tomography (PET) agent.

The study will also evaluate the patient safety and radiation safety of the EnLightTM, and the safety for the device operators and surgical staff of the LightPathTM Imaging System.

DETAILED DESCRIPTION:
This is a pilot study that is prospective, open-label, single-centre in nature in patients with gastric, pancreas, bile duct or duodenal cancer in whom tumour excision surgery is indicated.

Patients who give written informed consent will be screened for the study (Visit 1). Patients will undergo a positron emission tomography (PET) whole body scan. Screening assessments, including the PET scan, must be performed no less than 60 days before surgery and may be performed on the day of surgery.

On the day of surgery (Visit 2), subject's blood glucose level will be measured. Subjects with a blood glucose level < 12 mmol/l will receive an intravenous injection of 2-5 Mega Becquerel/kg (MBq/kg), up to a maximum 300 MBq of fluorine-18 fluorodeoxyglucose (18F-FDG) prior to surgery.

During surgery and not less than 120 minutes after injection of FDG, the primary lesion will be imaged using the EnLightTM system to determine margin status.

Gastrointestinal tumour excision surgery will then be performed according to standard of care. The surgical cavity and the lymph nodes will be imaged by the EnLightTM system to establish whether other radioactive tissue remain. These results will not influence any surgical or clinical decision-making, which will remain as standard of care. The resected tumour excision specimen will be imaged by the LightPathTM Imaging System. The resected tumour excision specimen will, in addition, be analysed according to standard of care pathology. The surgeon and surgical staff will be monitored for external exposure to ionizing radiation by means of dosimeters, and position sensors during surgery.

Patients will be followed-up (Visit 3) within a 2 - 14 day window after the end of surgery for adverse events (AEs). Those related to the use of the investigational devices, or the PET imaging agent will be identified as such.

ELIGIBILITY:
Inclusion Criteria:

1. Provides written informed consent to participate in the study.
2. Is a man or woman aged ≥ 30 years.
3. Patients diagnosed with gastric, pancreatic, bile duct or duodenal cancer whose treatment is to be tumour excision surgery.
4. Life expectancy of at least 12 months.
5. Blood glucose level < 12 mmol/l.

Exclusion Criteria:

1. Participation in another clinical study either concurrently or within 180 days prior to surgery.
2. Major surgery within 30 days before the baseline visit.
3. Women who are pregnant or lactating.
4. Renal impairment, hepatic impairment, serious infection or other life-threatening illness, other than cancer, within 60 days before surgery.
5. Previous exposure to ionizing radiation >5 millisieverts (mSv) in the previous 12 months.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female or male patients aged ≥ 30 years diagnosed with gastric, pancreatic, bile duct or duodenal cancer, whose treatment is to be tumour excision surgery.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
The location of PET imaging agent as measured by beta particle detection | Intraoperatively (during the single session of surgery on Day 0)
  The EnLightTM will be used for determining the number of lesions, their location and margin status, in the surgical cavity including within surrounding tissue, and lymph nodes. The EnLightTM is a beta particle detector used for imaging the location of the PET imaging agent. It works both in a hot-spot mode, to localise areas with high beta particle detection signal from the PET imaging agent, and in an imaging mode that allows video imaging of areas where the PET imaging agent has accumulated.
The location of PET imaging agent as measured by the LightPathTM Imaging System | Intraoperatively (during the single session of surgery on Day 0)
  The LightPathTM Imaging System will be used for determining the margin status of lesions and the metastatic involvement of lymph nodes.

SECONDARY OUTCOMES:
The number of lesions by histopathology | Expected on average Day 10 after surgery
  Number of lesions according to standard of care histopathology.
The number of metastatic lymph nodes by histopathology | Expected on average Day 10 after surgery
  The number of metastatic lymph nodes according to standard of care histopathology.
The extent of resection margins by histopathology | Expected on average Day 10 after surgery
  Extent of resection margins according to standard of care histopathology.
Ease of use measured by questionnaire | At the end of imaging on Day 0
  Ease of use measured by study-specific questionnaire
Radiation exposure | At the time of discharge to the ward after surgery on Day 0
  Radiological dose in microsieverts as measured by dosimeters worn by operating room staff
Number of participants with adverse events | Visit 3, at day 3-15
  Patients will be followed-up until Visit 3, 2-14 days after the end of surgery on Day 0 for adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl O'Farrell, PhD, Study Director — Head of Clinical Development
Locations (1):
- Semmelweis University First Clinic of Surgery, Budapest, Budapest, Hungary

REFERENCES:
- See also: Sponsor company's clinical trials website — http://www.lightpointmedical.com/clinical-trials/